CLINICAL TRIAL: NCT01892852
Title: Acupuncture Therapy for Chemotherapy-induced Peripheral Neuropathy in Lymphoma or Multiple Myeloma Patients: a Pilot Study
Brief Title: Acupuncture for Chemotherapy-induced Peripheral Neuropathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pusan National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AcuCIPN
Record Dates: First submitted 2013-06-18; First posted 2013-07-04 (Estimated); Last update posted 2013-07-17 (Estimated); Status verified 2013-07

CONDITIONS: Peripheral Neuropathy; Toxicity Due to Chemotherapy; Lymphoma; Multiple Myeloma
Keywords: Acupuncture; Traditional Korean Medicine
MeSH Terms: conditions — Peripheral Nervous System Diseases; Lymphoma; Multiple Myeloma | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acupuncture (Experimental): Acupuncture treatment
  Interventions: Procedure: Acupuncture
- Control (No Intervention): No other active treatment or sham acupuncture for this symptoms

INTERVENTIONS:
Procedure: Acupuncture — Acupuncture treatment will be performed by licensed doctors in Traditional Korean Medicine using 0.20 mm (diameter) X 0.40 mm (length) sized disposable acupuncture 3 times per week for 3 weeks. Acupuncture points are GV20, GB20 (bilateral), LI11 (bilateral), LI10 (bilateral), EX-UE9 (bilateral), ST36 (bilateral), ST40 (bilateral), and EX-LE10 (bilateral). Each session lasts 20-30 minutes.
  Arms: Acupuncture

SUMMARY:
The purpose of this study is to evaluate whether acupuncture can be effective for chemotherapy-induced peripheral neuropathy in lymphoma or multiple myeloma patients.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age and have diagnosis of a lymphoma or multiple myeloma.
* Patients must have chemotherapy-induced peripheral neuropathy greater or equal to 2 according to CTCAE (Common Terminology Criteria for Adverse Events) v 3.0 scale (Appendix A) in spite of previous conventional medications, e.g. Neurontin, Cymbalta and/or Lyrica. Patients receiving any of conventional medication for this symptoms must remain on the same medications throughout the study period.
* Patients, or the legal guardians of patients, must have the ability to understand Korean, and be ble to provide informed consent.
* ECOG (Eastern Cooperative Oncology Group) Performance Status of 0, 1, or 2.
* If the patient is a woman of child-bearing potential, she must have a negative urine pregnancy test and agree to use contraception.

Exclusion Criteria:

* Other diseases that, in the opinion of the investigators, can cause peripheral neuropathy, such as alcoholism, diabetes mellitus, and HIV.
* Current active treatment for lymphoma or multiple myeloma
* Ongoing local infection at or near the acupuncture point adopted in this trial.
* Severe immunocompromised patients, leukopenia ( < 4,000/㎣) or neutropenia ( < 1,500/㎣)
* Known coagulopathy, thrombocytopenia (< 50,000/㎣), and taking heparin (including low molecular weight heparin) or Coumadin at any dose.
* Serious emotional or mental problems that precludes study entry.
* Mental and physical disability that precludes accurate acupuncture.
* Serious systemic diseases such as active infection, severe heart disease, uncontrolled hypertension and diabetes mellitus.
* Cardiac pacemaker.
* Pregnant or breastfeeding
* Acupuncture therapy within the previous 30 days
* Concurrent other complementary and alternative therapy such as herbal agents, high dose vitamins, and etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2013-06; Primary Completion 2014-04 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Change of NCIC-CTC (National Cancer Institute of Canada - Common Toxicity Criteria) 4.0 scale from baseline | At baseline, 1, 2, 3, and 7 wks from baseline

SECONDARY OUTCOMES:
Change of VAS (Visual Analogue Scale) from baseline | At baseline, 1, 2, 3, and 7 wks from baseline
Change of FACT/GOG-Ntx (Functional Assessment of Cancer Therapy/Gynecologic Oncology Group Neurotoxicity) from baseline | At baseline, 1, 2, 3, and 7 wks from baseline
Adverse events | From study enrollment to the last follow-up (up to 7 wks)

CONTACTS AND LOCATIONS:
Overall Officials: Ho-Jin Shin, PhD, Principal Investigator — Pusan National University Hospital
Locations (1):
- Department of Hematology-Oncology and Center for Integrative Medicine, Pusan National University Hospital, Busan, South Korea